CLINICAL TRIAL: NCT01581593
Title: Multicenter, Open-label, Historically Controlled, Phase III Study to Assess the Efficacy, Tolerability, Safety and Pharmacokinetics of Kedrion IVIG 10% in Adult and Pediatric Subjects With Primary Immunodeficiency (PID).
Brief Title: Efficacy and Safety Study of Kedrion IVIG 10% to Treat Subjects With Primary Immunodeficiency (PID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kedrion S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB052
Record Dates: First submitted 2012-04-16; First posted 2012-04-20 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Primary Immunodeficiency; Agammaglobulinemia; Hypogammaglobulinemia; Antibody Deficiency
Keywords: Primary Immunodeficiency; PID; Agammaglobulinemia; Hypogammaglobulinemia; Antibody deficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Agammaglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kedrion IVIG 10% (Experimental): Kedrion IVIG 10% treatment.
  Interventions: Biological: Kedrion IVIG 10%

INTERVENTIONS:
Biological: Kedrion IVIG 10% — Dosage form - Intravenous (IV) infusion of Kedrion IVIG 10%; Dosage - 300 to 900 mg/kg body weight (bw); Frequency - every 21 to 28 days; Treatment duration - 12 months

SUMMARY:
The purpose of this study is to determine whether Kedrion IVIG 10% (an immunoglobulin solution) is effective in treating Primary Immunodeficiency (PID).

DETAILED DESCRIPTION:
People with primary immunodeficiency diseases (PID) have a defective immune system and experience recurrent protozoal, bacterial, fungal and viral infections. Antibody deficiencies make up the largest group of PIDs.

The standard care for patients with PID is replacement immunoglobulin (a class of antibodies) solution. Prophylactic treatment with intravenous immunoglobulin (IVIG) solution has been shown to increase the time free from serious infection.

Kedrion IVIG 10% is a new preparation of an immunoglobulin G (IgG) solution. Kedrion IVIG 10% will be given by IV infusion to all study participants. The data collected will help determine whether Kedrion IVIG 10% is suitable for treating PID subjects.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of a Primary Immunodeficiency Disease
* Male or female, ages 2 to 70 years
* Received 300-900 mg/kg of a licensed IVIG therapy at 21 or 28 day intervals for at least 3 months prior to this study
* 2 documented IgG trough levels of ≥ 5 g/L are obtained at two infusion cycles (21 or 28 days) within 12 months (one must be within 6 months) prior to study enrolment
* Non-pregnant females of child-bearing potential who agree to use adequate birth control during the study
* Subject is willing to comply with the protocol
* Authorization to access personal health information.
* Signed the informed consent form and a child assent form, if appropriate.
* If currently participating in a clinical trial with another experimental IVIG may be enrolled if they have received stable IVIG therapy for at least 3 infusion cycles prior to receiving Kedrion IVIG 10% and all inclusion and exclusion criteria are satisfied
* If currently participating in a trial of SCIG can be enrolled if they are switched to IVIG for three infusion cycles (21 or 28 days) prior to enrolment in this study

Exclusion Criteria:

* Has secondary immunodeficiency.
* Newly diagnosed and has not been treated with immunoglobulin or has been diagnosed with dysgammaglobulinemia or isolated IgG subclass deficiency.
* Has a history of repeated reactions or hypersensitivity to IVIG or other injectable forms of IgG.
* Has a history of thrombotic events defined by at least 1 event in subject's lifetime.
* Has IgA deficiency and is known to have antibodies to IgA.
* Has received blood products other than human albumin or human immunoglobulin within 12 months prior to enrolment.
* Has significant protein losing enteropathy, nephrotic syndrome or lymphangiectasia.
* Has an acute infection as documented by culture or diagnostic imaging and/or a body temperature exceeding 38.5 °C (101.3 °F) within 7 days prior to screening
* Has a known history or is positive at enrolment for human immunodeficiency virus (HIV) type 1 by NAT, hepatitis B virus (HBsAg and NAT), hepatitis C virus (by NAT), or hepatitis A virus (by NAT).
* Has levels of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times of the upper limit of normal for the laboratory designated for the study.
* Has an implanted venous access device
* Has profound anemia or persistent severe neutropenia (≤ 1000 neutrophils per mm3)or lymphopenia of less than 500 cells per microliter.
* Has a severe chronic condition such as renal failure (creatinine concentration > 2.0 times the upper limit of normal) with proteinuria, congestive heart failure (New York Heart Association III/IV), cardiomyopathy, cardiac arrhythmia associated with thromboembolic events (e.g. atrial fibrillation), unstable or advanced ischemic heart disease, hyperviscosity, or any other condition that the investigator believes is likely to interfere with evaluation of the study drug or with satisfactory conduct of the trial.
* Has a history of a malignant disease other than properly treated carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin within 24 months prior to enrolment.
* Has history of epilepsy or multiple episodes of migraine (defined as at least one episode within 6 months of enrolment) not completely controlled by medication.
* Is receiving steroids (oral or parenteral daily dose of ≥ 0.15 mg/kg/day of prednisone or equivalent) OR other immunosuppressive drugs or chemotherapy.
* Females who are pregnant, breast feeding or planning a pregnancy during the course of the study. Women who become pregnant during the study will be withdrawn from the study.
* Has participated in another clinical study within 3 weeks prior to study enrolment.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-11-12 (Actual); Primary Completion 2014-08-27 (Actual); Study Completion 2014-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mirella Calcinai, MD, Study Director — Kedrion SpA
Locations (15):
- United States (12):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Family Allergy & Asthma Center, PC, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Midwest Immunology Clinic, Plymouth, Minnesota
  - AAIR Research Center, Rochester, New York
  - Optimed Research, LTD, Columbus, Ohio
  - Dallas Allergy Immunology Research, Dallas, Texas
  - AARA Research Center, Dallas, Texas
  - Virginia Commonwealth University Health Systems, Richmond, Virginia
  - Marycliff Allergy Specialists, Spokane, Washington
- Canada (3):
  - Gordon Sussman Clinical Research Inc., Toronto, Ontario
  - Pediatric & Adult Allergy & Clinical Immunology, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Kedrion IVIG 10% 21 and 28 Days Infusion Schedule: Kedrion IVIG 10% treatment 21 and 28-day infusion schedule
  Kedrion IVIG 10%: Dosage form - Intravenous (IV) infusion of Kedrion IVIG 10%; Dosage - 300 to 900 mg/kg body weight (bw); Frequency - every 21 or 28 days; Duration - 12 months
Period: Overall Study
Arm/Group | Kedrion IVIG 10% 21 and 28 Days Infusion Schedule
Started | 45
Completed | 44
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Kedrion IVIG 10% 21 and 28 Day Infusion Schedule: Kedrion IVIG 10% 21 and 28 Day infusion schedule
  Kedrion IVIG 10%: Dosage form - Intravenous (IV) infusion of Kedrion IVIG 10%; Dosage - 300 to 900 mg/kg body weight (bw); Frequency - every 21 or 28 days; Treatment duration - 12 months
Arm/Group | Kedrion IVIG 10% 21 and 28 Day Infusion Schedule
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 27
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (20.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute, Serious Bacterial Infections in the Total ITT Population.
Description: The incidence of acute serious bacterial infections, e.g. bacterial pneumonia, bacteremia/sepsis, bacterial meningitis, visceral abscess, osteomyelitis/septic arthritis, meeting EMA and FDA criteria.
Time Frame: 13 months
Measure: Number (99% Confidence Interval); unit: ASBI's/person-year
Arm/Group | Kedrion IVIG 10% 21 and 28 Days Infusion Schedule
Number analyzed (Participants) | 45
ASBI's/person-year | 0.04 [0.00 to 0.11]

2. Secondary Outcome: Infections Other Than Acute, Serious Bacterial Infections (ASBIs) in the Total ITT Population.
Time Frame: 13 months
Measure: Number; unit: infect./subject's study duration (years)
Groups:
- Kedrion IVIG 10% 21 and 28 Days Infusion Schedule: Kedrion IVIG 10% treatment 21 and 28-day infusion schedule
  Kedrion IVIG 10%: Dosage form - Intravenous (IV) infusion of Kedrion IVIG 10%; Dosage - 300 to 900 mg/kg body weight (bw); Frequency - every 21 or 28 days; Treatment duration - 12 months
Arm/Group | Kedrion IVIG 10% 21 and 28 Days Infusion Schedule
Number analyzed (Participants) | 45
infect./subject's study duration (years)
  Upper respiratory tract infection | 0.42
  Sinusitis | 0.48
  Viral upper respiratory tract infection | 0.15
  Bronchitis | 0.11
  Nasopharyngitis | 0.11
  Rhinitis | 0.11
  Acute sinusitis | 0.15
  Gastroenteritis viral | 0.09
  Herpes zoster | 0.11
  Urinary tract infection | 0.11

3. Secondary Outcome: Days Out of Work/School/Daycare Due to Infection in the Total ITT Population.
Time Frame: 13 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- Kedrion IVIG 10% 21 & 28 Days Treatment Schedule: Kedrion IVIG 10% treatment.
  Kedrion IVIG 10%: Dosage form - Intravenous (IV) infusion of Kedrion IVIG 10%; Dosage - 300 to 900 mg/kg body weight (bw); Frequency - every 21 to 28 days; Treatment duration - 12 months
Arm/Group | Kedrion IVIG 10% 21 & 28 Days Treatment Schedule
Number analyzed (Participants) | 45
days | 2.8 (6.56)

4. Secondary Outcome: Days Unable to Perform Normal Daily Activities Due to Infection in the Total ITT Population.
Time Frame: 13 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kedrion IVIG 10% 21 and 28 Days Infusion Schedule
Number analyzed (Participants) | 45
days | 3.4 (6.53)

5. Secondary Outcome: Days on Therapeutic Antibiotics in the Total ITT Population.
Time Frame: 13 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kedrion IVIG 10% 21 and 28 Days Infusion Schedule
Number analyzed (Participants) | 45
days | 23.3 (33.77)

6. Secondary Outcome: Days of Unscheduled Visits to Physicians in the Total ITT Population.
Time Frame: 13 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kedrion IVIG 10% 21 and 28 Days Infusion Schedule
Number analyzed (Participants) | 45
days | 0.9 (1.14)

7. Secondary Outcome: Number of Hospitalizations Due to Infection in ITT Population.
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Kedrion IVIG 10% 21 & 28 Days Treatment Schedule
Number analyzed (Participants) | 45
Participants
  0 hospitalizations | 42
  1 hospitalization | 2
  2 hospitalizations | 1
  ≥ 3 hospitalizations | 0

8. Secondary Outcome: Days of Hospitalization Due to Infection in the Total ITT Population.
Time Frame: 13 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- Kedrion IVIG 10% 21 & 28 Days Treatments Schedule: Kedrion IVIG 10% treatment.
  Kedrion IVIG 10%: Dosage form - Intravenous (IV) infusion of Kedrion IVIG 10%; Dosage - 300 to 900 mg/kg body weight (bw); Frequency - every 21 to 28 days; Treatment duration - 12 months
Arm/Group | Kedrion IVIG 10% 21 & 28 Days Treatments Schedule
Number analyzed (Participants) | 45
days | 0.6 (2.21)

9. Secondary Outcome: Yearly Hospitalization Rate Due to Infection in the Total ITT Population.
Time Frame: 13 months
Measure: Mean (Standard Deviation); unit: hospitalizations per year
Arm/Group | Kedrion IVIG 10% 21 & 28 Days Treatments Schedule
Number analyzed (Participants) | 45
hospitalizations per year | 0.11 (0.436)

10. Secondary Outcome: Yearly Hospitalization Duration Due to Infection in the Total ITT Population.
Time Frame: 13 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kedrion IVIG 10% 21 & 28 Days Treatments Schedule
Number analyzed (Participants) | 45
days | 0.55 (2.196)

11. Secondary Outcome: Distribution of All-cause Hospitalizations in the Total ITT Population.
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Groups:
- Kedrion IVIG 10% 21 and 28 Days Treatment Schedule: Kedrion IVIG 10% treatment.
  Kedrion IVIG 10%: Dosage form - Intravenous (IV) infusion of Kedrion IVIG 10%; Dosage - 300 to 900 mg/kg body weight (bw); Frequency - every 21 to 28 days; Treatment duration - 12 months
Arm/Group | Kedrion IVIG 10% 21 and 28 Days Treatment Schedule
Number analyzed (Participants) | 45
Participants
  0 hospitalizations | 41
  1 hospitalization | 1
  2 hospitalizations | 2
  3 hospitalizations | 1
  ≥ 4 hospitalizations | 0

12. Secondary Outcome: Duration of All-cause Hospitalizations
Time Frame: 13 months
Population: The duration of the hospitalizations was measured for each of four subjects who were hospitalized and was calculated dividing by the subject's study duration in days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kedrion IVIG 10% 21 and 28 Days Treatment Schedule
Number analyzed (Participants) | 4
days | 17.8 (12.07)

13. Secondary Outcome: Distribution of Fever Episodes in the Total ITT Population.
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Kedrion IVIG 10% 21 and 28 Days Treatment Schedule
Number analyzed (Participants) | 45
Participants
  0 fever episodes | 34
  1 fever episode | 6
  2 fever episodes | 2
  3 fever episodes | 1
  4 fever episodes | 1
  5 fever episodes | 1

14. Secondary Outcome: Duration of Fever Episodes
Time Frame: 13 months
Population: The duration of fever episodes was measured for each of eleven subjects who experienced this event.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kedrion IVIG 10% 21 and 28 Days Treatment Schedule
Number analyzed (Participants) | 11
days | 6.5 (4.87)

15. Secondary Outcome: IgG Trough Levels at Steady State in the Total ITT Population.
Time Frame: 13 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Kedrion IVIG 10% 21 and 28 Days Treatment Schedule
Number analyzed (Participants) | 45
mg/dL | 888 (197)

ADVERSE EVENTS:
Time Frame: 13 months
Groups:
- Kedrion IVIG 10%: Kedrion IVIG 10% treatment.
  Kedrion IVIG 10%: Dosage form - Intravenous (IV) infusion of Kedrion IVIG 10%; Dosage - 300 to 900 mg/kg body weight (bw); Frequency - every 21 to 28 days; Duration - 12 months
Arm/Group | Kedrion IVIG 10%
Serious Adverse Events (participants affected / at risk) | 4/45
Other Adverse Events (participants affected / at risk) | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kedrion IVIG 10% (N=45)
Bacterial pneumonia (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kedrion IVIG 10% (N=45)
Upper Respiratory Tract Infection (Infections and infestations) | 13 (18)
Sinusitis (Infections and infestations) | 11 (22)
Viral Upper Respiratory Infection (Infections and infestations) | 5 (7)
Rhinitis (Infections and infestations) | 4 (5)
Acute Sinusitis (Infections and infestations) | 3 (6)
Bronchitis (Infections and infestations) | 3 (3)
Gastroenteritis Viral (Infections and infestations) | 3 (4)
Nasopharyngitis (Infections and infestations) | 3 (4)
Urinary Tract Infection (Infections and infestations) | 3 (5)
Pyrexia (General disorders) | 11 (22)
Fatigue (General disorders) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (19)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Adverse drug reaction (General disorders) | 3 (3)
Headache (Nervous system disorders) | 12 (21)
Sinus Headache (Nervous system disorders) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 8 (12)
Nausea (Gastrointestinal disorders) | 4 (7)
Vomiting (Gastrointestinal disorders) | 4 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Investigations (Investigations) | 12 (21)
Insomnia (Psychiatric disorders) | 4 (4)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 6 (18)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3)
Eye Disorders (Eye disorders) | 4 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (5)
Immune System Disorders (Immune system disorders) | 3 (4)
Vascular Disorders (Vascular disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No